CLINICAL TRIAL: NCT02648542
Title: The Effects of Compensatory Auditory Stimulation and Transcranial Direct Current Stimulation on Tinnitus Perception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soterix Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CASTDCS001
Record Dates: First submitted 2015-12-30; First posted 2016-01-07 (Estimated); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Transcranial Direct Current Stimulation; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CAS vs. tDCS (Active Comparator): Assess the efficacy of compensatory auditory stimulation (CAS) versus transcranial direct current stimulation (tDCS)
  Interventions: Other: Compensatory auditory stimulation; Device: transcranial direct current stimulation
- Combined CAS+tDCS vs. Sham (Sham Comparator): Assess the efficacy of combined compensatory auditory stimulation (CAS) + transcranial direct current stimulation (tDCS) versus sham stimulation
  Interventions: Other: Combined CAS and tDCS; Other: Sham stimulation

INTERVENTIONS:
Other: Compensatory auditory stimulation — Compensating for peripheral hearing loss by adjusting sound levels based on individual audiogram.
  Other Names: CAS
  Arms: CAS vs. tDCS
Device: transcranial direct current stimulation — Low-current electrical brain stimulation
  Other Names: tDCS
  Arms: CAS vs. tDCS
Other: Combined CAS and tDCS — Combined auditory and electrical stimulation
  Other Names: CAS + tDCS
  Arms: Combined CAS+tDCS vs. Sham
Other: Sham stimulation — Sham stimulation
  Other Names: Sham
  Arms: Combined CAS+tDCS vs. Sham

SUMMARY:
This study evaluates the ability of compensatory auditory stimulation (CAS) and transcranial direct current stimulation (tDCS) to help alleviate tinnitus. Subjects will receive CAS, tDCS, and the combination of the two to assess the effectiveness of the treatment.

DETAILED DESCRIPTION:
Tinnitus refers to persistent "ringing in the ears" in absence of external sound. For some individuals tinnitus can be disabling. Most tinnitus is of idiopathic origin and currently there are no reliable treatment options available. Existing approaches, such as hearing aids, counseling, and noise masking typically provide only partial relief and only for a minority of patients. Newer exploratory methods include tailored auditory stimulation and various brain stimulation techniques. While these techniques show great promise in a subset of subjects (maybe about 1/3), it is hard to anticipate which, if any, will benefit a given patient.

Transcranial Direct Current Stimulation (tDCS) has been explored for a number of neurological conditions, and it is most effective when paired with some form of training (e.g. motor rehab after stroke). For tinnitus however this treatment modality has only been tested in isolation. The purpose of this pilot study is to explore the benefits of combining tailored compensatory auditory stimulation with tDCS.

There is widespread consensus in the research community that tinnitus originates with some peripheral hearing deficit, and that maladaptive central plastic mechanisms subsequently lead to the tinnitus percept. Most individuals with tinnitus have audiometric evidence of hearing loss. Our hypothesis is that reduced input to the auditory pathway leads to increased sensitivity (auditory gain) and finally aberrant activity in the frequency band with hearing loss. In this view, auditory stimulation that compensates for the reduced input can potentially revert the maladaptive plasticity.This is consistent with the reported benefits of hearing aids and tailored auditory stimulation. Our hypothesis is that tDCS can boost adaptation induced by compensatory auditory stimulation to reduce the strength of the phantom percept.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-80 years of age
* No history of otological disease
* Subjects with hearing loss, hyperacusis and/or tinnitus are eligible to participate

Exclusion Criteria:

* hearing loss greater than 50 dB HL
* Shows signs of depression or anxiety (Zung self-rating Depression Scale > 50; Beck Anxiety Inventory > 36)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Reduction in minimum masking levels | 2 weeks
  Measurement of the minimum masking level required to mask the subjective tinnitus loudness is assessed after each intervention.
Reduction in tinnitus percept as assessed via the visual analog test of tinnitus loudness | 2 weeks
  Measurement of the subjective loudness of the tinnitus percept is measured using the visual analog scale test after each intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Lucas C Parra, Ph.D., Principal Investigator — City College of New York, CUNY

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared if requested